CLINICAL TRIAL: NCT01297439
Title: CONTRADYS : A Randomized Controlled Trial of a New Prophylactic Maneuver, the "Pushing" Maneuver, Aiming to Reduce the Risk for Shoulder Dystocia
Brief Title: New Prophylactic Maneuver: the "Pushing" Maneuver, Aiming to Reduce the Risk for Shoulder Dystocia
Acronym: CONTRADYS
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: the study stopped due to the lack of inclusion.
Sponsor: Assistance Publique - Hôpitaux de Paris (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: P091109
Record Dates: First submitted 2011-02-09; First posted 2011-02-16 (Estimated); Last update posted 2015-04-30 (Estimated); Status verified 2015-04

CONDITIONS: Shoulder Dystocia,; Brachial Plexus Injury; Asphyxia,; Hematoma,; Clavicle Fracture,; Humerus Fracture.
Keywords: shoulder dystocia,; Mac Roberts' maneuver,; pushing maneuver
MeSH Terms: conditions — Shoulder Dystocia; Asphyxia; Hematoma; Humeral Fractures

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No

ARMS (2):
- group M (Other): Normal delivery without "pushing" maneuver suctioning of fetal nose and mouth during delivery
  Interventions: Procedure: suctioning of fetal nose and mouth during delivery
- group C (Experimental): "Pushing" maneuver on the fetal head
  Interventions: Procedure: Pushing maneuver

INTERVENTIONS:
Procedure: suctioning of fetal nose and mouth during delivery — Normal delivery without "pushing" maneuver: either an expectative attitude or a suctioning of fetal nose and mouth during delivery, since the crowning of the head (appearance of the fetal scalp at the introitus between pushes).
  Other Names: M:Mouchage meaning suctioning of fetal nose and mouth
  Arms: group M
Procedure: Pushing maneuver — The "pushing" maneuver is performed gently on the fetal head since the crowning of the head (appearance of the fetal scalp at the introitus between pushes), during one uterine contraction, aiming to facilitate the anterior shoulder to slip off behind the symphysis pubis, reducing thus the risk of shoulder dystocia.
  Other Names: C ;"contre pulsion" in French, meaning "Pushing maneuver"
  Arms: group C

SUMMARY:
Shoulder dystocia is a major obstetric emergency defined as a delivery requiring maneuver in addition to downward traction on the fetal head for delivery of the shoulders. Shoulder dystocia is a major obstetrical complication, occurring in approximately 0.2 to 3% of deliveries, principally due to fetal macrosomia. The obstetrical and neonatal complications associated with shoulder dystocia include newborn mortality occurring in 21 to 290 per 1000 deliveries, generalized asphyxia, fractures, neurological damages (brachial plexus injury) and hematoma. The objective of this study was to evaluate the "pushing" maneuver, that is performed gently on the fetal head since the crowning of the head (appearance of the fetal scalp at the introitus between pushes), aiming to facilitate the anterior shoulder to slip off behind the symphysis pubis, reducing thus the risk of shoulder dystocia. This preventive maneuver may reduce the power (energy/time unit) exerted on the perineal tissues and give the shoulders time to enter the pelvic cavity. The "pushing" maneuver will be evaluated in comparison with either an expectative attitude or a suctioning of fetal nose and mouth.

DETAILED DESCRIPTION:
Hypothesis: the "pushing" maneuver reduces of 50% the risk of shoulder dystocia in comparison with either an expectative attitude or a suctioning of fetal nose and mouth.

Main objective: to assess whether prophylactic use of the "pushing on the fetal head" maneuver decreases the prevalence of shoulder dystocia, in comparison with an expectative attitude or a suctioning of fetal nose and mouth.

Secondary objective: to compare the occurrence of neonatal complications including brachial plexus injury, clavicle and humerus fracture, hematoma and generalized asphyxia.

Main criterion: occurrence of shoulder dystocia, defined by a necessity of requiring a specific obstetrical maneuver (McRoberts' maneuver).

Secondary criterion: neonatal complications including neurological damages (brachial plexus injury), generalized asphyxia, hematoma, clavicle and humerus fractures.

Methods: prospective, randomized, multicenter blind study with a modified intention-to-treat analysis. Patients are included during the last obstetrical consultation and randomized in the delivery room.

Number of patients (α error, β error): a sample size of 1126 patients was calculated to allow detection of a 50% reduction of shoulder dystocia, with a prevalence of dystocia reaching 4.3% in usual deliveries (expectative attitude or suctioning of fetal nose and mouth), with a 65% dystocia risk decrease in the group C (α error of 0.05, β error of 0.20).

Inclusion and exclusion criteria. Inclusion: women having completed 37 or more gestational weeks with singleton vertex fetus, delivering vaginally. Exclusion: patients with caesarean section are excluded.

Place of the study: department of gynecology and obstetrics, BEAUJON hospital, Clichy, France and department of gynecology and obstetrics, BICHAT hospital, Paris, France.

Duration of inclusion: two years and 6 months Duration of patients' participation: two months maximum Duration of the study: two years and 9 months. Mean number of inclusion each month: 30 Number of investigation centre: 2 (BEAUJON hospital, BICHAT hospital).

ELIGIBILITY:
Inclusion Criteria:

* women having completed 37 or more gestational weeks with singleton vertex fetus, delivering vaginally

Exclusion Criteria:

* patients with caesarean section are excluded

Ages: 18 Years to 45 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 1538 (Actual)
Dates: Start 2011-03; Primary Completion 2013-11 (Actual); Study Completion 2014-03 (Actual)

PRIMARY OUTCOMES:
occurrence of shoulder dystocia | during delivery
  shoulder dystocia is defined as a necessity of requiring a specific obstetrical maneuver (McRoberts' maneuver).

SECONDARY OUTCOMES:
complications | 5 days after delivery
  neonatal complications including neurological damages (brachial plexus injury), generalized asphyxia, hematoma, clavicle and humerus fractures.

CONTACTS AND LOCATIONS:
Overall Officials: Olivier Poujade, MD, Principal Investigator — Assistance Publique Hopitaux de Paris
Locations (1):
- Hôpital Beaujon, Clichy, France